CLINICAL TRIAL: NCT00522197
Title: A Phase II Trial of ACAPHA in Former Smokers With Intraepithelial Neoplasia
Brief Title: ACAPHA in Preventing Lung Cancer in Former Smokers With Bronchial Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000562055; U01CA096109 (NIH); BCCA-H02-61177-A002; BCCA-R02-1177
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; small cell lung cancer; squamous lung dysplasia
MeSH Terms: conditions — Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — antitumor A; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACAPHA (Active Comparator)
  Interventions: Dietary Supplement: multi-herbal agent ACAPHA
- Sugar Pill (Placebo Comparator)
  Interventions: Dietary Supplement: Sugar Pill

INTERVENTIONS:
Dietary Supplement: multi-herbal agent ACAPHA
  Arms: ACAPHA
Dietary Supplement: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of ACAPHA, a combination of six herbs, may prevent lung cancer from forming in former smokers with bronchial intraepithelial neoplasia.

PURPOSE: This randomized phase II trial is studying the side effects and how well ACAPHA works in preventing lung cancer in former smokers with bronchial intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of multi-herbal agent ACAPHA in former smokers with bronchial intraepithelial neoplasia.
* Evaluate whether ACAPHA can modulate other surrogate endpoint biomarkers of aberrant methylation, cell cycle regulation, apoptosis, as well as phase I and II enzyme regulation.
* Establish a library of in vivo confocal microendoscopy images with corresponding histopathology, nuclear morphometry, and other biomarker information to assess the potential of confocal microendoscopy as a nonbiopsy method in assessing the effect of chemoprevention agents.

OUTLINE: Patients are stratified according to gender. Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral multi-herbal agent ACAPHA twice daily for 6 months. Patients achieving a partial response receive an additional 6 months of ACAPHA.
* Arm II: Patients receive oral placebo twice daily for 6 months. Patients achieving a partial response receive an additional 6 months of placebo. Patients with progressive disease receive ACAPHA twice daily for 6 months.

Patients undergo sputum cytology, oral and bronchial brushings, bronchoalveolar lavage, and bronchial tissue biopsies at baseline and at 6 and 12 months. Samples are analyzed for histopathological and morphometric cell changes; MIB-1 bcl-2, and TUNEL immunostaining; methylation biomarkers; and gene expression analysis of RNA.

After completion of study therapy, patients are followed at 1 and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One or more areas of bronchial intraepithelial neoplasia (IEN) (metaplasia/dysplasia) with a nuclear morphometry index > 1.36 and a surface diameter > 1.2 mm on autofluorescence bronchoscopy
* Atypical sputum cells as determined by computer-assisted image analysis
* Former smoker (i.e., stopped smoking at least 1 year ago) who has smoked at least 30 pack-years (i.e., 1 pack/day for 30 years or more)
* Exhaled carbon monoxide level < 5 ppm
* No invasive cancer on bronchoscopy or abnormal spiral chest CT scan suspicious of lung cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0 or 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Normal renal function tests (BUN, creatinine, urinalysis)
* Normal liver function tests (AST, ALT, bilirubin, alkaline phosphatase)
* No chronic active hepatitis or liver cirrhosis
* No acute bronchitis or pneumonia within the past month
* No known reaction to xylocaine
* No medical condition that, in the opinion of the investigator, could jeopardize the patient's safety during participation in the study, including any of the following:

  * Acute or chronic respiratory failure
  * Unstable angina
  * Uncontrolled congestive heart failure
  * Bleeding disorder

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-09; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of multi-herbal agent ACAPHA as measured by combined histopathology and nuclear morphometry of intraepithelial neoplasia lesions | 12 months

SECONDARY OUTCOMES:
Changes in the severity of dysplasia by bronchial biopsy | 6 months
Changes in the morphometric index of sputum cells, bronchial biopsies, and epithelial cells in the bronchoalveolar lavage fluid (BAL) | 12 months
MIB-1, bcl-2, and TUNEL immunostaining in the bronchial biopsies | 12 months
Methylation biomarkers in the sputa, oral brush, and BAL cells | 12 months
Gene expression analysis of RNA from bronchial brush cells | 12 months
Volumetric measurement of CT scan-detected lung nodules before and after treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Principal Investigator — British Columbia Cancer Agency